CLINICAL TRIAL: NCT06959329
Title: The Influence of Intensified Sensory Stimulation on Upper Extremity Sensory Parameters and Motor Function in Children With Developmental Coordination Disorder
Brief Title: Influence of Sensory Stimulation on Sensory Parameters and Motor Function in Children With Developmental Coordination Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Collaborators: Daugavpils University, Department of Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAR/2025/mar/01
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Developmental Coordination Disorder
Keywords: developmental coordination disorder; sensory function; motor function; sensory stimulation; adolescents
MeSH Terms: conditions — Motor Skills Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statisticians responible for data processing and analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard therapy without intensified tactile stimulation (Active Comparator): Intervention: Passive and active therapy without high sensory stimulation Duration: 4 weeks Frequency: 3 sessions per week Session duration: 60 minutes
  Intervention structure:
  Interventions: Other: Active and passive physical therapy without intensified sensory stimulation
- Therapy with intensified tactile stimulation (Experimental): Intervention: Passive and active therapy incorporating high sensory stimulation Duration: 4 weeks Frequency: 3 sessions per week Session duration: 60 minutes
  Interventions: Other: Active and passive physical therapy with intensified sensory stimulation

INTERVENTIONS:
Other: Active and passive physical therapy without intensified sensory stimulation — Intervention: Passive and active therapy without high sensory stimulation Duration: 4 weeks Frequency: 3 sessions per week Session duration: 60 minutes
  Intervention structure:
  Passive therapy (30 minutes):
  • Stroking and rubbing techniques from classic massage applied in the area of arm forearm and hand with low force and frequency upper limb massage - 15 minutes per limb
  Active therapy (30 minutes): upper limb muscle strengthening exercises (without globalized vibration); difficulty level individually adjusted to meet participants' current potential, so that in the last sets/reps little manual assistance from the therapist is needed:
  * Supine pull-ups - 3 sets of 8 reps, ~45 seconds rest between sets
  * Standing pull-ups - 3 sets of 8 reps, ~45 seconds rest between sets
  * Standing push-ups - 3 sets of 8 reps, ~45 seconds rest between sets
  * Standing elbow extensions - 3 sets of 8 reps, ~45 seconds rest between sets
  Arms: Standard therapy without intensified tactile stimulation
Other: Active and passive physical therapy with intensified sensory stimulation — Intervention: Passive and active therapy incorporating high sensory stimulation Duration: 4 weeks Frequency: 3 sessions per week Session duration: 60 minutes
  Intervention structure:
  Passive therapy (30 minutes): stimulation of joint receptors, muscle spindles, and tactile pathways:
  * High-frequency soft tissue mobilisations
  * Localised high-amplitude vibration (30-50 Hz; Galileo Mano 30, Novotec Medical GmbH)
  * Deep pressure techniques - Wilbarger brushing protocol followed by joint compressions Active therapy (30 minutes): upper limb and shoulder girdle muscle strengthening exercises with globalized vibration using Redcord Stimula (30-50 Hz; Redcord AS, Norway); difficulty level individually adjusted to meet participants' current potential. Excercises the same as in the control group.
  Arms: Therapy with intensified tactile stimulation

SUMMARY:
The goal of this clinical trial is to evaluate whether intensive sensory stimulation therapy can improve upper limb motor skills and sensory function in children aged 12-16 years with severe symptoms of Developmental Coordination Disorder (DCD). The main questions it aims to answer are:

1. Will children with DCD who undergo intensive sensory stimulation therapy show greater improvement in upper limb motor function compared to those receiving standard therapy?
2. Will intensive sensory stimulation therapy lead to better sensory function outcomes, including joint position sense, resistance sense, pressure sense, temperature perception, and two-point discrimination? Researchers will compare children receiving intensive sensory stimulation therapy to those receiving standard therapy without intensive sensory stimulation to see if the targeted intervention results in superior improvements in motor and sensory function.

DETAILED DESCRIPTION:
Background Developmental Coordination Disorder (DCD) is a neurodevelopmental condition that affects the development of motor skills in children, impacting their ability to perform a range of daily activities (Missiuna et al., 2008; Zwicker et al., 2012). According to the Diagnostic and Statistical Manual of Mental Disorders (American Psychiatric Association, 2013), DCD is characterized by difficulties in acquiring and executing coordinated movements.

The diagnostic criteria for DCD include motor abilities that are significantly below what would be expected for the individual's chronological age and learning experiences. These motor challenges must interfere substantially with daily living activities, educational or professional achievements, and hobbies. Symptoms typically emerge in early childhood and cannot be better explained by intellectual disability, neurological conditions affecting movement, or visual impairments. Motor difficulties often present as clumsiness, slowness, and inaccuracy in executing movements (Lachambre et al., 2021).

Recent research highlights the high prevalence and significant impact of sensory processing impairments among children with DCD. Studies have identified notable differences across various sensory domains - including visual, tactile, proprioceptive, auditory, and vestibular processing - when compared to typically developing peers (Tran et al., 2022). Children with DCD, for instance, exhibit greater deficits in proprioceptive processing, such as difficulties with localizing single and double simultaneous stimuli, graphesthesia, finger identification (Elbasan et al., 2012; Malloy-Miller et al., 1995), and two-point discrimination under both dynamic and static conditions (Law et al., 2011).

Children with DCD experience pronounced sensory differences that significantly affect their daily functioning. These sensory differences may also signal the presence of additional neurodivergent traits. Furthermore, sensory processing impairments are closely associated with poor motor coordination and have a substantial impact on daily activities (Keating et al., 2024).

Design and hypotheses The planned study is a randomised controlled trial (RCT) aimed at evaluating the effectiveness of intensive sensory stimulation therapy on upper limb motor skills and sensory function in children with pronounced symptoms of DCD, as assessed by The Movement Assessment Battery for Children - Second Edition (MABC-2).

Main hypotheses:

H1: Children with DCD who undergo intensive therapy involving sensory stimulation will show a significant improvement in upper limb motor function compared to children in the control group after four weeks of intervention.

H2: Children with DCD receiving intensive sensory stimulation will demonstrate significant improvements in upper extremity sensory function compared to the control group.

Specific hypotheses:

H2a: After four weeks of intensive sensory stimulation, children in the experimental group will exhibit better joint position sense compared to children in the control group.

H2b: After four weeks of intensive sensory stimulation, children in the experimental group will show an improved sense of resistance in the upper limb compared to the control group.

H2c: Children in the experimental group will demonstrate better temperature perception than those in the control group.

H2d: Children in the experimental group will display enhanced sense of pressure compared to the control group.

H2e: Children in the experimental group will demonstrate better two-point discrimination sense compared to children in the control group.

General procedure Participant Recruitment and Screening Children aged 12-16 with pronounced symptoms of DCD, identified using The Movement Assessment Battery for Children - Second Edition (MABC-2), will be recruited from the local clinics, schools, and rehabilitation centres.

Inclusion and exclusion criteria are described elsewhere in this record. The M-ABC-2 is a standardized tool used to assess motor coordination and identify movement difficulties in children aged 3 to 16 years. The test version for the age band 11-16 years wil be used. The test's tasks are grouped into three core domains: Manual Dexterity, Aiming and Catching, and Balance. Manual Dexterity tasks evaluate fine motor skills through activities like threading beads or placing pegs. Aiming and Catching tasks focus on hand-eye coordination using items like balls and beanbags. Balance tasks test both static and dynamic balance, such as standing on one leg or walking heel-to-toe along a straight line. The assessment typically takes about 20 minutes. Standardized instructions and materials are used to ensure consistency. Each task is scored based on the accuracy or time taken to complete it. These raw scores are then converted into standard scores and percentile ranks using normative data for the child's age group. Children with scores ranging from 40 to 50 standard points (=pronounced DCD symptoms) will be included.

Based on data from our previous research, we estimated that a total sample size of 82 participants (i.e., 41 per group) is required to achieve sufficient statistical power to detect meaningful differences between the groups. Given the anticipated length and demands of the intervention, we expect an attrition rate of approximately 15% due to potential dropouts. To account for this, we adjusted our recruitment target accordingly (total required N~94).

Baseline Assessment Before the intervention begins, all participants will undergo a baseline assessment. This will include: evaluation of upper limb motor skills using standardised motor tasks from the The Jebsen-Taylor Hand Function Test (JTHFT; Jebbsen et al., 1969; Fabbri et al., 2021); assessment of joint position sense, sense of resistance, sense of temperature, sense of pressure, and two-point discrimination sense.

The JTHFT is a standardized assessment designed to evaluate hand function in relation to everyday tasks. It is commonly used in rehabilitation and clinical settings to measure both fine and gross motor skills in individuals with neurological or musculoskeletal impairments, such as DCD. The test is appropriate for children over the age of five and provides normative data to allow comparison across age and gender groups. The JTHFT includes seven timed subtests, each simulating a daily activity involving the hands. These tasks are: writing a short sentence, turning over cards, picking up and placing small common objects, simulating feeding with a spoon, stacking checkers, moving light cans, and moving heavy cans. These subtests are performed individually, and each is timed in seconds, with shorter completion times indicating better hand function. The test is administered separately for each hand, typically beginning with the non-dominant hand, and it takes approximately 15 minutes.

To ensure consistency, the JTHFT is administered using a standardized protocol that includes specific instructions for each task, standardized materials, and defined starting positions.

Assessments will be conducted by trained evaluators who are blinded to group allocation.

Randomisation Participants will be randomly assigned to either: experimental group (with intensified sensory stimulation), or control group (without intensified sensory stimulation).

To ensure unbiased allocation of participants and equal group sizes, randomisation will be carried out using a computer-generated random number method. Participants will be randomised into either the experimental or control group using a simple randomisation method with allocation concealment, designed for continuous recruitment. Because the full list of participants is not available in advance, each participant will be randomised individually upon enrolment. To ensure equal group sizes over time, an adaptive control mechanism will be used once the halfway point of recruitment is approached. If a group begins to exceed its target number, subsequent participants will be automatically allocated to the underfilled group to maintain balance.

Intervention Phase (4 weeks) Experimental group: Participants will engage in a structured therapy programme focusing on intensive sensory stimulation of the upper limbs. Control group: Participants will receive an equivalent volume therapy programme without intensive sensory stimulation. Therapists administering interventions will follow a standardised protocol to ensure consistency (described esewhere in this record). All physiotherapists delivering the intervention in this study have undergone comprehensive training to ensure high-quality implementation of the intervention protocol. Prior to the start of the study, each physiotherapist will complete a structured training program, including both theoretical instruction and practical application of all intervention components. Their competence will be verified through supervised practice sessions and fidelity assessments, during which they demonstrated a high level of proficiency and adherence to the protocol. The intervention procedures have been developed and refined based on previous experiences. All procedures are non-invasive and have been designed to minimise any physical or psychological burden on participants. While participants may experience temporary fatigue, particularly during physical activity components, no significant risks are anticipated. The physiotherapists are trained to monitor participants closely throughout the intervention sessions and to respond appropriately to any signs of distress or adverse events.

Post-Intervention Assessment Immediately after completing the 4-week intervention, all participants will undergo a second assessment identical to the baseline assessment.

Evaluators will again be blinded to group assignments to minimise bias. Data Analysis Statistical analysis will compare pre- and post-intervention results between the experimental and control groups. Differences in motor performance and sensory function outcomes will be analysed using appropriate statistical tests (e.g., repeated-measures ANOVA, t-tests, non-parametric statistics), depending on data distribution.

Ethical Considerations The study protocol will be approved by an appropriate Research Ethics Committee. All procedures will adhere to ethical standards for research involving human participants, including confidentiality, the right to withdraw, and risk minimisation.

Outcome measures All outcome measures are described in detail elsewhere in this record. All assessors conducting the outcome measurements have undergone rigorous training and demonstrated excellent proficiency in administering the assessment tools. All outcome measures utilised in this study have been previously tested in pilot studies across diverse participant groups and have shown reliability ranging from good to excellent, with intraclass correlation coefficients (ICC) exceeding 0.8. All procedures employed in the study are considered safe. Participants may experience only minimal discomfort during certain assessments, such as pressure sensation testing. However, no significant risks are anticipated. The study protocol has been designed to prioritise participant safety and to ensure that any potential discomfort is transient and within ethically acceptable limits.

ELIGIBILITY:
Inclusion Criteria:

* between 12-16 years of age
* diagnosed severe symptoms of the developmental coordination disorder based on The Movement Assessment Battery for Children 2nd Edition (M-ABC 2), with scores ranging from 40 to 50
* typical intellectual development (i.e., children attending mainstream education)
* voluntary participation and informed consent signed by parents or legal guardians

Exclusion Criteria:

* current or previous diagnosis of serious orthopaedic or neurological conditions (e.g. fractures, congenital deformities, cerebral palsy, etc.)
* history of any surgical procedures
* history of significant musculoskeletal pain or dysfunction lasting more than two weeks and requiring medical or physiotherapeutic intervention, or any such symptoms occurring within one month prior to the study
* any current musculoskeletal dysfunction and/or pain
* body mass index exceeding 22 kg/m³

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The Jebsen-Taylor Hand Function Test (JTHFT) | From enrollment to the end of treatment at 4 weeks
  The JTHFT (Jebsen et al. 1969, Fabbri et al. 2021) is a standardized assessment tool used to evaluate the hand function of individuals, particularly in clinical settings. This test is particularly relevant for assessing fine motor skills and the ability to perform tasks that require both coordination and dexterity.
  The tasks include:
  Writing a Sentence: Assesses the ability to hold a pen and write legibly. Turning Over Cards: Tests finger dexterity by flipping a set of cards one at a time.
  Picking Up Small Objects: Evaluates the ability to manipulate small items, often using a pre-defined set of objects.
  Simulated Feeding: Involves using utensils to demonstrate the ability to eat. Stacking Checkers: Measures the manipulation of objects by stacking them. Lifting a Paper Clip: Assesses fine motor skills by picking up a small, light object.
Joint Position Sense | From enrollment to the end of treatment at 4 weeks
  Joint position sense is assessed using active reproduction and position differentiation tests. In reproduction, the participant memorises a target position (90º shoulder abduction) and then attempts to replicate it without visual input. In differentiation, they aim to reach half the target angle (45º). An electronic inclinometer (±1º accuracy) fixed to the upper arm measures angles. Markers are placed on anatomical landmarks, and a goniometer is secured parallel to the humeral axis. Tests are performed seated. The target position is passively assumed under supervision and memorised (×3). The participant then reproduces or differentiates the angle (×2 each), confirming with "stop." Readings are taken after each attempt. Both sides are tested. The absolute positioning error (absolute difference between target and assumed angles) is used for analysis, based on the mean of two measurements.
Sense of Resistance | From enrollment to the end of treatment at 4 weeks
  Resistance sense is assessed using force reproduction and differentiation tests. In the first, the participant replicates a memorised reference force; in the second, they generate half that force. An electronic dynamometer (±0.1 kG accuracy) is attached to a 12 cm sleeve on the upper arm and connected to the floor via an elastic cord. Tests are conducted in 90º shoulder flexion or abduction. The reference force is defined as the effort needed to stretch the elastic cord slightly for 5 seconds. After adjustments, this is repeated three times, and the participant memorises the force. Then, with eyes closed, they reproduce or halve the force, confirming with "stop." The examiner records the values. Each test is repeated three times. Two extremities are tested. The absolute force generation error (normalised difference in %) is used for analysis, based on the mean of three measurements.
Sense of Pressure | From enrollment to the end of treatment at 4 weeks
  Pressure sense is assessed at 5 fixed points on the chest, upper limb, and scapular region, corresponding to different peripheral nerve branches. The test is performed in supine or prone position, depending on the site, with the upper limb abducted to 90º. An algometer is used to apply focused pressure and record force. It has a blunt tip with a 20 mm² contact area and measures with ±0.1 kG accuracy. During testing (eyes closed), the participant says "stop" when pressure at a point becomes uncomfortable but not painful. The examiner records the force at that moment. Each point is tested twice. Pressure is applied perpendicularly to the skin, and both sides are assessed. The maximum applied force does not exceed 6 kG to avoid subcutaneous bruising. The final result is the average of the two measurements.
Discriminative Sense | From enrollment to the end of treatment at 4 weeks
  Discriminative sense is tested at 5 fixed points on the chest, upper limb, and scapular area - same as in the pressure sense test. A calliper with two rounded tips is used, with a measurement accuracy of 0.5 mm. With the participant's eyes closed, the examiner applies both tips to the skin and gradually reduces the distance between them. The participant reports whether they feel one or two touch points. When they begin to perceive only one while two are still applied, the distance is recorded. This is repeated twice. The calliper arms are held perpendicular to the skin without added pressure - only the instrument's own weight acts on the surface. One arm always remains at a fixed point, while the other approaches from the side or from distal direction, depending on the location. Both sides of the body are tested. The final result is the average of the two measurements.
Sense of Temperature | From enrollment to the end of treatment at 4 weeks
  Temperature sense is assessed at 5 fixed points on the chest, upper limb, and scapular area, as in the pressure test. A custom-built device with a 3 cm² flat thermal head, heat converter, and digital thermometer is used, offering ±0.5ºC accuracy and precise heat control. With eyes closed, the participant detects a change in temperature. The test begins with the head at neutral temperature (30ºC), increasing steadily at 1ºC every 10 seconds. The participant says "stop" when they notice a temperature change, and the examiner records the reading. Each point is tested twice. A tolerance test is performed beforehand to define each participant's discomfort threshold. The stimulus never exceeds 45ºC. Both sides of the body are assessed. The final result is the average of the two measurements.

CONTACTS AND LOCATIONS:
Locations (2):
- Daugavpils University, Daugavpils, Latvia
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Because of the international character of the project, legal considerations may be an issue. If this is not the case, the data may be available on request.

REFERENCES:
- [Background] Keating J, Purcell C, Gerson SA, Vanderwert RE, Jones CRG. Exploring the presence and impact of sensory differences in children with Developmental Coordination Disorder. Res Dev Disabil. 2024 May;148:104714. doi: 10.1016/j.ridd.2024.104714. Epub 2024 Mar 13. PMID 38484422
- [Background] Law SH, Lo SK, Chow S, Cheing GL. Grip force control is dependent on task constraints in children with and without developmental coordination disorder. Int J Rehabil Res. 2011 Jun;34(2):93-9. doi: 10.1097/MRR.0b013e32833f0519. PMID 21178635
- [Background] Elbasan B, Kayihan H, Duzgun I. Sensory integration and activities of daily living in children with developmental coordination disorder. Ital J Pediatr. 2012 Apr 30;38:14. doi: 10.1186/1824-7288-38-14. PMID 22546072
- [Background] Tran HT, Li YC, Lin HY, Lee SD, Wang PJ. Sensory Processing Impairments in Children with Developmental Coordination Disorder. Children (Basel). 2022 Sep 22;9(10):1443. doi: 10.3390/children9101443. PMID 36291382
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.). Arlington: American Psychiatric Publishing, 2013.
- [Background] Lachambre C, Proteau-Lemieux M, Lepage JF, Bussieres EL, Lippe S. Attentional and executive functions in children and adolescents with developmental coordination disorder and the influence of comorbid disorders: A systematic review of the literature. PLoS One. 2021 Jun 4;16(6):e0252043. doi: 10.1371/journal.pone.0252043. eCollection 2021. PMID 34086687
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Developmental coordination disorder: a review and update. Eur J Paediatr Neurol. 2012 Nov;16(6):573-81. doi: 10.1016/j.ejpn.2012.05.005. Epub 2012 Jun 15. PMID 22705270
- [Background] Missiuna C, Gaines R, McLean J, Delaat D, Egan M, Soucie H. Description of children identified by physicians as having developmental coordination disorder. Dev Med Child Neurol. 2008 Nov;50(11):839-44. doi: 10.1111/j.1469-8749.2008.03140.x. Epub 2008 Sep 22. PMID 18811713
- [Background] Fabbri B, Berardi A, Tofani M, Panuccio F, Ruotolo I, Sellitto G, Galeoto G. A systematic review of the psychometric properties of the Jebsen-Taylor Hand Function Test (JTHFT). Hand Surg Rehabil. 2021 Oct;40(5):560-567. doi: 10.1016/j.hansur.2021.05.004. Epub 2021 May 21. PMID 34023565
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487